CLINICAL TRIAL: NCT06348238
Title: Strategies to Improve Well-Being and Diabetes Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Scharnetzki (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Scharnetzki, Faculty Scientist I, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2074997
Record Dates: First submitted 2024-03-04; First posted 2024-04-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are masked to their assigned condition until the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Affirmation (Experimental): Participants review a list of values and are instructed to choose up to two that are important to them. The values listed are intentionally unrelated to the threat-inducing domain so that the exercise broadens participants' focus. Next, participants are asked to write a few sentences about why their chosen values are important to them and identify times in which these values have helped them navigate challenges.
  Interventions: Behavioral: Self-Affirmation
- Waitlist Control (Sham Comparator): Participants in the waitlist control condition will also complete writing exercises but they will be abbreviated (this in the psychological literature is referred to as a "low affirmation condition"). At the end of the study, waitlist control participants will have access to the full exercise should they like to receive it.
  Interventions: Behavioral: Self-Affirmation

INTERVENTIONS:
Behavioral: Self-Affirmation — Self-affirmation theory contends that integrity of one's self-concept (self integrity) is essential for navigating daily stressors. When individuals encounter information or contexts that pose a threat to one's self-integrity, we can adopt maladaptive coping strategies to alleviate the discomfort. One strategy for strengthening self-integrity is engage in an explicit process of reinforcing sources of self-worth - self-affirmation. Self affirmation interventions have participants engage in an exercise writing about core personal values (a writing induction). In a writing induction, participants review a list of values and are instructed to choose up to two that are important to them. Participants are then asked to write a few sentences about why their chosen values are important to them and identify times in which these values have helped them navigate challenges.

SUMMARY:
This project aims to implement an adapted self-affirmation intervention among a population of individuals with diabetes to reduce the negative psychosocial impacts of stigma. In a self-affirmation, participants are guiding through a writing exercise writing designed to reinforce sources of self-worth before they encounter or engage in stressful or stigmatizing events. Participants in this study will be asked to complete self-affirmation exercises before their 3-month wellness appointments with their endocrinologists over the course of a year. The main questions the investigators are asking are:

* Will self-affirmation reduce feelings of stigmatization?
* Will self-affirmation increase self-efficacy and motivation to engage in condition management behaviors.
* Will self-affirmation improve blood glucose control. Participants will be randomly assigned to either the intervention condition or a waitlist control condition. Participants in the waitlist control condition will also complete writing exercises but they will be abbreviated (this in the psychological literature is referred to as a "low affirmation condition"). At the end of the study, waitlist control participants will have access to the full exercise should they like to receive it.

After each appointment and self-affirmation, participants will complete surveys assessing feelings of stigma and motivation to engage in condition management. All participants will already be using continuous glucose monitors. The investigators will compare both survey responses and continuous glucose data between our conditions to assess the efficacy of the self-affirmation intervention.

DETAILED DESCRIPTION:
Upon enrollment, participants will receive an electronic link to an enrollment survey to assess their baseline perceptions of diabetes and weight-based stigma, attitudes towards and intentions to engage in condition management behaviors, sociodemographic and clinical factors (e.g., gender, age, race, and ethnicity) and potential moderators, including diabetes distress, anxiety, depression, history of weight-based victimization, and stigma consciousness. Participants will then be randomly assigned to either the self-affirmation intervention or a waitlist control condition (participants in the waitlist control will have the option to receive the same intervention as participants in the experimental condition at end of the study period). Participants will be using the randomization module in our online survey vendor, REDCap. This module allows researchers to program REDcap to automatically randomize participants in their study to one of the arms or conditions of their study. Before every 3-month wellness visit with their endocrinologist, participants will receive an electronic prompt to complete a self-affirmation writing induction. To complete the writing induction, participants will review a list of values and are instructed to choose up to two that are important to them. Next, participants are asked to write a few sentences about why their chosen values are important to them and identify times in which these values have helped them navigate challenges. Participants in the waitlist control condition will also complete writing exercises but they will be abbreviated (this in the psychological literature is referred to as a "low affirmation condition"). At the end of the study, waitlist control participants will have access to the full exercise should they like to receive it. After their 3-month wellness visit, participants will be sent an electronic link to the post-intervention survey. This will assess to assess their baseline perceptions of diabetes and weight-based stigma, attitudes towards and intentions to engage in condition management behaviors. In total, participants will complete 4 writing inductions and 4 post-evaluation surveys over the course of a year. In addition to writing inductions and survey data, aggregated data from participants' continuous glucose monitors will be collected throughout the study period to assess time spend in target glucose range. The investigators will also collect participants' most recent pre-and-post intervention Hemoglobin A1C (HbA1c) measurements via EHR data to assess longitudinal changes in glucose control. To evaluate the effectiveness of our intervention, the investigators will test whether mean scores in 1) post-intervention stigma and stigma-induced identity threat scores; 2) average confidence in and intentions to engage in condition management scores; and 3) average time spent in target glycemic target range significantly differ between conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age, have a type 2 diabetes (T2D) diagnosis, and currently use a continue glucose monitor as part of their condition management.
* Participants must be patients of MaineHealth Endocrinology and Diabetes, be at least 18 years of age, have a type 2 diabetes (T2D) diagnosis, and currently use a continue glucose monitor as part of their condition management (Dexcom, FreeStyle Libre).

Exclusion Criteria:

* Individuals under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Social Identity Threat Concerns (SITC) Scale - Adapted for Diabetes | Immediately after each intervention; completed 4 times over the course of a year
  Used to assess participants' concerns about experiencing diabetes-specific stigma-induced identity threat while receiving care for T2D. A 1 (Strongly disagree) to 7 (Strongly agree) Likert response scale is used for all items. A composite score is created by summing all items. Higher values indicate greater social identity threat concerns.
Social Identity Threat Concerns (SITC) Scale - Adapted for Weight | Immediately after each intervention; completed 4 times over the course of a year
  Used to assess participants' concerns about experiencing weight-specific stigma-induced identity threat while receiving care for T2D. A 1 (Strongly disagree) to 7 (Strongly agree) Likert response scale is used for all items. A composite score is created by summing all items. Higher values indicate greater social identity threat concerns.
Diabetes Stigma Assessment Scale | Immediately after each intervention; completed 4 times over the course of a year
  6-item subscale assessing participants perceived and experienced stigma for use with adults with diabetes. A 1(strongly disagree) to 5 (strongly agree) Likert response scale is used for all items. A composite score is created by summing all items. Higher values indicate greater diabetes stigma.
Diabetes Stigma Assessment Scale - Adapted for weight stigma | Immediately after each intervention; completed 4 times over the course of a year
  6-item subscale assessing participants perceived and experienced stigma for use with adults with diabetes. We adapted this measure to anchor on internalized weight stigma. A 1(strongly disagree) to 5 (strongly agree) Likert response scale is used for all items. A composite score is created by summing all items. Higher values indicate greater diabetes stigma.
The Revised Diabetes Self-Management Questionnaire | Immediately after each intervention; completed 4 times over the course of a year
  27-items measure to assess uptake of essential self-management practices for Diabetes. A 0 (Does not apply to me) to 3 (Applies to me very much) Likert response scale is used for all items.
Confidence in Diabetes Self-Care Scale | Immediately after each intervention; completed 4 times over the course of a year
  20-item measure assessing patient self-efficacy, confidence in ability to perform diabetes self-care tasks. A 1 ("No, I am sure I cannot") to 5 ("Yes, I am sure I can") Likert response scale is used for all items. A composite score is created by summing all items. Higher values indicate greater confidence.
Blood glucose | Through study completion, an average of 1 year
  Continuous glucose monitor derived indices for time spent in-range

SECONDARY OUTCOMES:
Hemoglobin A1C | Collected once at time of study enrollment and once at study completion
  Blood assay assessing average blood glucose level; Will be collected as part of EPIC data requests; HbA1c will be requested at the time of study enrollment and throughout study completion (5 total)
Patient-reported age | at end of study (1 year)
  Patient's self-reported age in years
Patient Gender | Collected once at time of study enrollment
  Patient's self-reported gender identity; They may select as many as apply from the following: Man, Woman, Transgender, Gender Queer/Gender non-conforming, Non-Binary, Different Identity (Please specify), Prefer not to answer
Patient Race | Collected once at time of study enrollment
  Patient's self-reported racial identity. They may select as many as apply from the following: White, Black, Asian, Native American or Alaska Native, Middle Eastern or North African, Native Hawaiian or other Pacific Islander Different Identity(Please specify) Prefer not to answer
Patient ethnicity | Collected once at time of study enrollment
  Patient's self-reported ethnicity: Are you of Hispanic, Latino or Spanish origin, such as Mexican, Puerto Rican, or Cuban? Yes, No, Prefer not to answer
Patient's highest level of education completed | Collected once at time of study enrollment
  Patient's self-reported highest level of education completed; They may select from:
  8th grade or less, Some high school, High school diploma/GED, Some college or technical school classes, no degree, Associate's or Bachelor's degree, Master's, doctorate, or professional degree, Prefer not to answer
Household income | Collected once at time of study enrollment
  Patient's self-reported household income: Which of the following categories best describes the total income for the household where you live?
  * Less than $20,000
  * Between $20,000 and $70,000
  * More than $70,000
  * Don't know/Not sure
  * Prefer not to answer
Zip code | Collected once at time of study enrollment
  Patients will be asked to provide a value for the following question: What is the zip code for the area where you currently live? Zip codes will be converted to Rural-Urban Commuting Area Codes, which are used to classify census tracts into rural and urban categories.
Years since diagnosis | Collected once at time of study enrollment
  Patients' will provide a value for the following question: How many years has it been since you were first diagnosed with Type 2 Diabetes?
  Diabetes diagnosis and year of diabetes diagnosis will also be verified as part of an EPIC data request
Diabetes Management Plan | Collected once at time of study enrollment
  Patients' will provide a value for the following question: Which of the following options best describes how you manage your Type 2 Diabetes?
  * Diet
  * Medication
  * Both diet and medication
  If Medication or Both diet and medication is selected:
  Please tell us more about medications and medication dosages you are currently taking to manage your diabetes: ______________________
Physical activity | Collected once at time of study enrollment
  Patients' will provide text responses for the following questions:
  What kind of physical activity do you do? How often do you do this activity (days per week) How long do you typically do this activity for (minutes)
Continuous glucose monitor use | Collected once at time of study enrollment
  Patients' will provide a value for the following question:
  How long have you been using your continuous glucose monitor (in months or years)?
Height | Collected once at time of study enrollment
  Patient's height (feet and inches) will be collected as part of an EPIC data request; this will be used to calculate BMI
Weight | Collected once at time of study enrollment
  Patient's weight (pounds) will be collected as part of an EPIC data request; this will be used to calculate BMI
History of weight-based victimization (moderator/covariate) | Collected once at time of study enrollment
  3-item measure assessing experiences of weight-based discrimination. A binary Yes/No response scale is used for all items. The number of affirmative responses will be summed to create a composite. Higher scores indicate greater weight-based victimization.
Problem Areas in Diabetes Questionnaire (moderator/covariate) | Collected once at time of study enrollment
  20-item measure of diabetes-related emotional distress that assesses a broad range of feelings related to living with diabetes. A 0 (Not a problem) to 4 (Serious problem) Likert response scale is used for all items. A composite score is created by summing all items. Higher values indicate greater distress.
Generalized Anxiety Disorder 7-item (moderator/covariate) | Collected once at time of study enrollment
  7-item measure of generalized anxiety disorder. A 0 (Not at all) to 3 (Nearly every day) Likert response scale is used for all items. A composite score is created by summing all items. Higher values indicate greater anxiety.
Patient Health Questionnaire (PHQ-9) (moderator/covariate) | Collected once at time of study enrollment
  9-item measure of depression severity. A 0 (Not at all) to 3 (Nearly every day) Likert response scale is used for all items. A composite score is created by summing all items. Higher values indicate greater depression.
Stigma Consciousness Questionnaire (moderator/covariate) | Collected once at time of study enrollment
  10-item measure to predict the degree to which stigmatized groups expect to be stereotyped and discriminated against by others. These items will be adapted to measure stigma consciousness relating to diabetes and health care. A 0 (strongly disagree) to 6(strongly agree) Likert scale, with a midpoint of 3 (neither agree nor disagree) is used for all items. A composite score is created by summing all items. Higher values indicate greater stigma consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Scharnetzki, Principal Investigator — MaineHealth
Locations (1):
- MaineHealth Institute for Research, Center for Interdisciplinary and Population Health Research, Westbrook, Maine, United States

IPD SHARING:
Plan to Share IPD: Yes
Our findings will be shared with the science and local communities through scientific publications and professional conference presentations. To ensure study findings are reproduceable, per best practice, statistical code for our analyses will be made available on open science platforms (e.g., Open Science Framework), and deidentified, aggregated data may be available upon request by members of the scientific community. All findings will be reported at the group-level, so nothing can be tied to participants as individuals.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Upon completion of data collection and throughout the publication and dissemination period.

REFERENCES:
- [Background] Bayer R. Stigma and the ethics of public health: not can we but should we. Soc Sci Med. 2008 Aug;67(3):463-72. doi: 10.1016/j.socscimed.2008.03.017. Epub 2008 May 24. PMID 18502551
- [Background] Centers for Disease Control and Prevention. (2002). About Prediabetes & Type 2 Diabetes. Retrieved from https://www.cdc.gov/diabetes/prevention/about-prediabetes.html
- [Background] Puhl RM, Heuer CA. Obesity stigma: important considerations for public health. Am J Public Health. 2010 Jun;100(6):1019-28. doi: 10.2105/AJPH.2009.159491. Epub 2010 Jan 14. PMID 20075322
- [Background] Major, B., Hunger, J. M., Bunyan, D. P., & Miller, C. T. (2014). The ironic effects of weight stigma. Journal of Experimental Social Psychology, 51, 74-80. https://doi.org/10.1016/j.jesp.2013.11.009
- [Background] Wu YK, Berry DC. Impact of weight stigma on physiological and psychological health outcomes for overweight and obese adults: A systematic review. J Adv Nurs. 2018 May;74(5):1030-1042. doi: 10.1111/jan.13511. Epub 2017 Dec 8. PMID 29171076
- [Background] Vadiveloo M, Mattei J. Perceived Weight Discrimination and 10-Year Risk of Allostatic Load Among US Adults. Ann Behav Med. 2017 Feb;51(1):94-104. doi: 10.1007/s12160-016-9831-7. PMID 27553775
- [Background] Talumaa B, Brown A, Batterham RL, Kalea AZ. Effective strategies in ending weight stigma in healthcare. Obes Rev. 2022 Oct;23(10):e13494. doi: 10.1111/obr.13494. Epub 2022 Aug 7. PMID 35934011
- [Background] Himmelstein MS, Puhl RM. At multiple fronts: Diabetes stigma and weight stigma in adults with type 2 diabetes. Diabet Med. 2021 Jan;38(1):e14387. doi: 10.1111/dme.14387. Epub 2020 Sep 23. PMID 32799378
- [Background] Steele, C. M. (1988). The psychology of self-affirmation: Sustaining the integrity of the self. In L. Berkowitz (Ed.), Advances in experimental social psychology, Vol. 21. Social psychological studies of the self: Perspectives and programs (pp. 261-302). Academic Press.
- [Background] Epton T, Harris PR. Self-affirmation promotes health behavior change. Health Psychol. 2008 Nov;27(6):746-52. doi: 10.1037/0278-6133.27.6.746. PMID 19025270
- [Background] Armitage CJ, Harris PR, Hepton G, Napper L. Self-affirmation increases acceptance of health-risk information among UK adult smokers with low socioeconomic status. Psychol Addict Behav. 2008 Mar;22(1):88-95. doi: 10.1037/0893-164X.22.1.88. PMID 18298234
- [Background] Sherman, D. A., Nelson, L. D., & Steele, C. M. (2000). Do messages about health risks threaten the self? Increasing the acceptance of threatening health messages via self-affirmation. Personality and Social Psychology Bulletin, 26(9), 1046-1058.
- [Background] Cohen GL, Sherman DK. The psychology of change: self-affirmation and social psychological intervention. Annu Rev Psychol. 2014;65:333-71. doi: 10.1146/annurev-psych-010213-115137. PMID 24405362
- [Background] Centers for Disease Control and Prevention (2022, June 29). National Diabetes Statistics Report Estimates of Diabetes and Its Burden in the United States. Retrieved April 8, 2023, from https://www.cdc.gov/diabetes/data/statistics-report/index.html
- [Background] American Diabetes Association (2022, July 28). Statistics About Diabetes. Retrieved April 8, 2023, from https://diabetes.org/about-us/statistics/about-diabetes#:~:text=Prevalence%20in%20seniors%3A%20The%20percentage,diagnosed%20with%20diabetes%20every%20year.
- [Background] Hoyt CL, Burnette JL, Thomas FN, Orvidas K. Public Health Messages and Weight-Related Beliefs: Implications for Well-Being and Stigma. Front Psychol. 2019 Dec 17;10:2806. doi: 10.3389/fpsyg.2019.02806. eCollection 2019. PMID 31920849
- [Background] Major B, O'Brien LT. The social psychology of stigma. Annu Rev Psychol. 2005;56:393-421. doi: 10.1146/annurev.psych.56.091103.070137. PMID 15709941
- [Background] Puhl RM, Himmelstein MS, Hateley-Browne JL, Speight J. Weight stigma and diabetes stigma in U.S. adults with type 2 diabetes: Associations with diabetes self-care behaviors and perceptions of health care. Diabetes Res Clin Pract. 2020 Oct;168:108387. doi: 10.1016/j.diabres.2020.108387. Epub 2020 Aug 26. PMID 32858100
- [Background] Saguy AC, Frederick D, Gruys K. Reporting risk, producing prejudice: how news reporting on obesity shapes attitudes about health risk, policy, and prejudice. Soc Sci Med. 2014 Jun;111:125-33. doi: 10.1016/j.socscimed.2014.03.026. Epub 2014 Mar 28. PMID 24785268
- [Background] Lee KM, Hunger JM, Tomiyama AJ. Weight stigma and health behaviors: evidence from the Eating in America Study. Int J Obes (Lond). 2021 Jul;45(7):1499-1509. doi: 10.1038/s41366-021-00814-5. Epub 2021 May 1. PMID 33934109
- [Background] Schabert J, Browne JL, Mosely K, Speight J. Social stigma in diabetes : a framework to understand a growing problem for an increasing epidemic. Patient. 2013;6(1):1-10. doi: 10.1007/s40271-012-0001-0. PMID 23322536
- [Background] Steele, C. M., Spencer, S. J., & Aronson, J. (2002). Contending with group image: The psychology of stereotype and social identity threat. In M. P. Zanna (Ed.), Advances in experimental social psychology, Vol. 34, pp. 379-440). Academic Press. https://doi.org/10.1016/S0065-2601(02)80009-0
- [Background] Hunger JM, Major B, Blodorn A, Miller CT. Weighed down by stigma: How weight-based social identity threat contributes to weight gain and poor health. Soc Personal Psychol Compass. 2015 Jun;9(6):255-268. doi: 10.1111/spc3.12172. Epub 2015 Jun 4. PMID 29225670
- [Background] Shapiro JR, Neuberg SL. From stereotype threat to stereotype threats: implications of a multi-threat framework for causes, moderators, mediators, consequences, and interventions. Pers Soc Psychol Rev. 2007 May;11(2):107-30. doi: 10.1177/1088868306294790. PMID 18453458
- [Background] Shapiro JR. Different groups, different threats: a multi-threat approach to the experience of stereotype threats. Pers Soc Psychol Bull. 2011 Apr;37(4):464-80. doi: 10.1177/0146167211398140. PMID 21441217
- [Background] Steele CM. A threat in the air. How stereotypes shape intellectual identity and performance. Am Psychol. 1997 Jun;52(6):613-29. doi: 10.1037//0003-066x.52.6.613. PMID 9174398
- [Background] Schmader T, Johns M, Forbes C. An integrated process model of stereotype threat effects on performance. Psychol Rev. 2008 Apr;115(2):336-56. doi: 10.1037/0033-295X.115.2.336. PMID 18426293
- [Background] Muraven M, Baumeister RF. Self-regulation and depletion of limited resources: does self-control resemble a muscle? Psychol Bull. 2000 Mar;126(2):247-59. doi: 10.1037/0033-2909.126.2.247. PMID 10748642
- [Background] Polonsky WH, Fisher L, Guzman S, Villa-Caballero L, Edelman SV. Psychological insulin resistance in patients with type 2 diabetes: the scope of the problem. Diabetes Care. 2005 Oct;28(10):2543-5. doi: 10.2337/diacare.28.10.2543. No abstract available. PMID 16186296
- [Background] Ritholz MD, Smaldone A, Lee J, Castillo A, Wolpert H, Weinger K. Perceptions of psychosocial factors and the insulin pump. Diabetes Care. 2007 Mar;30(3):549-54. doi: 10.2337/dc06-1755. PMID 17327319
- [Background] Sherman, D. A. K., Nelson, L. D., & Steele, C. M. (2000). Do messages about health risks threaten the self? Increasing the acceptance of threatening health messages via self-affirmation. Personality and Social Psychology Bulletin, 26(9), 1046-1058. https://doi.org/10.1177/01461672002611003
- [Background] Sherman, D. K., Lokhande, M., Müller, T., & Cohen, G. L. (2021). Self affirmation interventions. In G. M. Walton & A. J. Crum (Eds.), Handbook of wise interventions: How social psychology can help people change (pp. 63-99). The Guilford Press.
- [Background] Sherman, D. K., & Cohen, G. L. (2006). The psychology of self-defense: Self-affirmation theory. In M. P. Zanna (Ed.), Advances in experimental social psychology, Vol. 38, pp. 183-242). Elsevier Academic Press. https://doi.org/10.1016/S0065-2601(06)38004-5
- [Background] Ferrer RA, Cohen GL. Reconceptualizing Self-Affirmation With the Trigger and Channel Framework: Lessons From the Health Domain. Pers Soc Psychol Rev. 2019 Aug;23(3):285-304. doi: 10.1177/1088868318797036. Epub 2018 Oct 7. PMID 30295141
- [Background] Epton T, Harris PR, Kane R, van Koningsbruggen GM, Sheeran P. The impact of self-affirmation on health-behavior change: a meta-analysis. Health Psychol. 2015 Mar;34(3):187-96. doi: 10.1037/hea0000116. Epub 2014 Aug 18. PMID 25133846
- [Background] Sherman DK, Hartson KA, Binning KR, Purdie-Vaughns V, Garcia J, Taborsky-Barba S, Tomassetti S, Nussbaum AD, Cohen GL. Deflecting the trajectory and changing the narrative: how self-affirmation affects academic performance and motivation under identity threat. J Pers Soc Psychol. 2013 Apr;104(4):591-618. doi: 10.1037/a0031495. Epub 2013 Feb 11. PMID 23397969
- [Background] Cohen GL, Garcia J, Apfel N, Master A. Reducing the racial achievement gap: a social-psychological intervention. Science. 2006 Sep 1;313(5791):1307-10. doi: 10.1126/science.1128317. PMID 16946074
- [Background] Cohen GL, Garcia J, Purdie-Vaughns V, Apfel N, Brzustoski P. Recursive processes in self-affirmation: intervening to close the minority achievement gap. Science. 2009 Apr 17;324(5925):400-3. doi: 10.1126/science.1170769. PMID 19372432
- [Background] Miyake A, Kost-Smith LE, Finkelstein ND, Pollock SJ, Cohen GL, Ito TA. Reducing the gender achievement gap in college science: a classroom study of values affirmation. Science. 2010 Nov 26;330(6008):1234-7. doi: 10.1126/science.1195996. PMID 21109670
- [Background] Walton GM, Cohen GL. A brief social-belonging intervention improves academic and health outcomes of minority students. Science. 2011 Mar 18;331(6023):1447-51. doi: 10.1126/science.1198364. PMID 21415354
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Cohen, J. (1988). Statistical Power Analysis for the Behavioral Sciences, 2nd Edn. New York, NY: Academic Press.
- [Background] Kang H. Sample size determination and power analysis using the G*Power software. J Educ Eval Health Prof. 2021;18:17. doi: 10.3352/jeehp.2021.18.17. Epub 2021 Jul 30. PMID 34325496
- [Background] Hatzenbuehler ML, Phelan JC, Link BG. Stigma as a fundamental cause of population health inequalities. Am J Public Health. 2013 May;103(5):813-21. doi: 10.2105/AJPH.2012.301069. Epub 2013 Mar 14. PMID 23488505
- [Background] Stangl AL, Earnshaw VA, Logie CH, van Brakel W, C Simbayi L, Barre I, Dovidio JF. The Health Stigma and Discrimination Framework: a global, crosscutting framework to inform research, intervention development, and policy on health-related stigmas. BMC Med. 2019 Feb 15;17(1):31. doi: 10.1186/s12916-019-1271-3. PMID 30764826
- [Background] Meadows A, Higgs S. The Multifaceted Nature of Weight-Related Self-Stigma: Validation of the Two-Factor Weight Bias Internalization Scale (WBIS-2F). Front Psychol. 2019 Apr 16;10:808. doi: 10.3389/fpsyg.2019.00808. eCollection 2019. PMID 31040808
- [Background] Browne JL, Ventura AD, Mosely K, Speight J. Measuring the Stigma Surrounding Type 2 Diabetes: Development and Validation of the Type 2 Diabetes Stigma Assessment Scale (DSAS-2). Diabetes Care. 2016 Dec;39(12):2141-2148. doi: 10.2337/dc16-0117. Epub 2016 Aug 11. PMID 27515964
- [Background] Van Der Ven NC, Weinger K, Yi J, Pouwer F, Ader H, Van Der Ploeg HM, Snoek FJ. The confidence in diabetes self-care scale: psychometric properties of a new measure of diabetes-specific self-efficacy in Dutch and US patients with type 1 diabetes. Diabetes Care. 2003 Mar;26(3):713-8. doi: 10.2337/diacare.26.3.713. PMID 12610027
- [Background] Schmitt A, Kulzer B, Ehrmann D, Haak T, Hermanns N. A Self-Report Measure of Diabetes Self-Management for Type 1 and Type 2 Diabetes: The Diabetes Self-Management Questionnaire-Revised (DSMQ-R) - Clinimetric Evidence From Five Studies. Front Clin Diabetes Healthc. 2022 Jan 13;2:823046. doi: 10.3389/fcdhc.2021.823046. eCollection 2021. PMID 36994332
- [Background] Chehregosha H, Khamseh ME, Malek M, Hosseinpanah F, Ismail-Beigi F. A View Beyond HbA1c: Role of Continuous Glucose Monitoring. Diabetes Ther. 2019 Jun;10(3):853-863. doi: 10.1007/s13300-019-0619-1. Epub 2019 Apr 29. PMID 31037553
- [Background] Puhl RM, Latner JD, King KM, Luedicke J. Weight bias among professionals treating eating disorders: attitudes about treatment and perceived patient outcomes. Int J Eat Disord. 2014 Jan;47(1):65-75. doi: 10.1002/eat.22186. Epub 2013 Sep 5. PMID 24038385
- [Background] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Background] Pinel EC. Stigma consciousness: the psychological legacy of social stereotypes. J Pers Soc Psychol. 1999 Jan;76(1):114-28. doi: 10.1037//0022-3514.76.1.114. PMID 9972557
- [Background] Swinburn BA, Kraak VI, Allender S, Atkins VJ, Baker PI, Bogard JR, Brinsden H, Calvillo A, De Schutter O, Devarajan R, Ezzati M, Friel S, Goenka S, Hammond RA, Hastings G, Hawkes C, Herrero M, Hovmand PS, Howden M, Jaacks LM, Kapetanaki AB, Kasman M, Kuhnlein HV, Kumanyika SK, Larijani B, Lobstein T, Long MW, Matsudo VKR, Mills SDH, Morgan G, Morshed A, Nece PM, Pan A, Patterson DW, Sacks G, Shekar M, Simmons GL, Smit W, Tootee A, Vandevijvere S, Waterlander WE, Wolfenden L, Dietz WH. The Global Syndemic of Obesity, Undernutrition, and Climate Change: The Lancet Commission report. Lancet. 2019 Feb 23;393(10173):791-846. doi: 10.1016/S0140-6736(18)32822-8. Epub 2019 Jan 27. No abstract available. PMID 30700377
- [Background] Puhl RM, Himmelstein MS, Pearl RL. Weight stigma as a psychosocial contributor to obesity. Am Psychol. 2020 Feb-Mar;75(2):274-289. doi: 10.1037/amp0000538. PMID 32053000
- [Background] Liu NF, Brown AS, Folias AE, Younge MF, Guzman SJ, Close KL, Wood R. Stigma in People With Type 1 or Type 2 Diabetes. Clin Diabetes. 2017 Jan;35(1):27-34. doi: 10.2337/cd16-0020. PMID 28144043
- [Background] van Koningsbruggen GM, Das E. Don't derogate this message! Self-affirmation promotes online type 2 diabetes risk test taking. Psychol Health. 2009 Jul;24(6):635-49. doi: 10.1080/08870440802340156. PMID 20205017
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] American Psychological Association. (n.d.). APA Dictionary of Psychology. American Psychological Association. https://dictionary.apa.org/wait-list-control-group
- [Background] Kroeper, K. M., Williams, H. E., Thompson, S., Hernandez-Colmenares, A., Mills, A., Spencer, S. J., & Murphy, M. C. (in progress). The Social Identity Threat Concerns Scale [data analysis and writing ongoing].

DOCUMENTS (1):
  • Informed Consent Form (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT06348238/ICF_000.pdf